CLINICAL TRIAL: NCT03006796
Title: Observational Prospective stUdy of aZilsartan Medoxomil/ Chlorthalidone Compared With Irbesartan/hydrochlorothiaZide Combination Therapy in Patients With arteriaL Hypertension and obEsity in Routine Clinical Practice (PUZZLE).
Brief Title: Observational Study of Azilsartan/Chlorthalidone and Irbesartan/Hydrochlorothiazide in Hypertension and Obesity.
Acronym: PUZZLE
Status: Completed | Type: Observational
Sponsor: Russian Heart Failure Society (Other)
Responsible Party: Principal Investigator, Yury Vasyuk, professor, Russian Heart Failure Society
Other Study IDs: IISR-2015-101477
Record Dates: First submitted 2016-12-27; First posted 2016-12-30 (Estimated); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: Arterial Hypertension
Keywords: Obesity
MeSH Terms: conditions — Hypertension; Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- group 1 (AZL/C): Group 1 - patients receiving azilsartan medoxomil/chlorthalidone 40/12.5 mg or 40/25 mg per os once a day for 6 months.
- group 2 (IRB/H): Group 2 - patients receiving irbesartan/hydrochlorothiazide 150/12.5 mg or 300/25 mg per once a day for 6 months.

SUMMARY:
This is an observational prospective study of azilsartan medoxomil / chlorthalidone compared with irbesartan / hydrochlorothiazide in routine therapy of patients with arterial hypertension and obesity.

DETAILED DESCRIPTION:
Observational Prospective stUdy of aZilsartan medoxomil/ chlorthalidone compared with irbesartan/hydrochlorothiaZide combination therapy in patients with arteriaL hypertension and obEsity in routine clinical practice (PUZZLE).

The study population is 94 patients with untreated or poorly controlled arterial hypertension and obesity.

The main inclusion criteria are:

1. Male and female 35-55 year old.
2. Diagnosis of essential arterial hypertension I-II grade.
3. Patients with obesity (BMI ≥ 30 kg/m²)
4. Patients with untreated arterial hypertension (clinic SBP ≥ 140 mmHg, DBP ≥ 90 mmHg and no previous antihypertensive treatment.
5. Patients with poorly controlled arterial hypertension (clinic SBP ≥ 140 mmHg, DBP ≥ 90 mmHg on previous antihypertensive treatment.
6. Written informed consent.

The main exclusion criteria are:

1. Patients with symptomatic organ damage (myocardial infarction, stroke, angina pectoris, chronic kidney disease ≥ 4 grade, diabetes).
2. Patients with secondary arterial hypertension.
3. Patients with intolerance of angiotensin II receptor blockers, thiazide diuretic.
4. Patients with contraindication to study drugs in accordance with Russian instruction.
5. Patients currently enrolled in other clinical trials. The treatment period is 6 months. The study plan includes 4 basic and 1 additional visits are planned: initial visit, 3 follow-ups (including additional) and study-end visit.

ELIGIBILITY:
Inclusion Criteria:

1. male and female 35-55 year old,
2. diagnosis of I-II grade essential AH,
3. patients with obesity (BMI ≥ 30 kg/m²),
4. patients with untreated AH (office SBP ≥ 140 mmHg, DBP ≥ 90 mmHg, no previous antihypertensive therapy),
5. patients with poorly controlled AH (office SBP ≥ 140 mmHg, DBP ≥ 90 mmHg on previous antihypertensive therapy),
6. written informed consent form (ICF).

Exclusion Criteria:

1. patients with symptomatic organ damage (myocardial infarction, stroke, angina pectoris, chronic kidney disease stage ≥ 4, diabetes),
2. patients with intolerance of ARB, thiazide diuretics,
3. secondary AH,
4. patients with contraindication to study drugs in accordance with Russian instruction,
5. patients currently enrolled in other clinical trials.

Ages: 35 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: The study population is 94 patients with untreated or poorly controlled arterial hypertension and obesity 35-55 years old.
Sampling Method: Probability Sample
Enrollment: 94 (Actual)
Dates: Start 2017-01-16 (Actual); Primary Completion 2020-02 (Actual); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
Clinic systolic blood pressure lowering. | From baseline (Month 0) to the study-end visit (Month 6)
  Lowering of clinic systolic blood pressure.

SECONDARY OUTCOMES:
24-hour systolic brachial and central blood pressure lowering. | From baseline (Month 0) to the study-end visit (Month 6).
  Lowering of ambulatory brachial and central blood pressure.
24-hour aortic pulse wave velocity reduction. | From baseline (Month 0) to the study-end visit (Month 6).
  Lowering of ambulatory aortic pulse wave velocity.
change in proportion of patients with normal and abnormal LV geometry with assessment of LV mass index and relative wall thickness. | From baseline (Month 0) to the study-end visit (Month 6).
  Normalization of abnormal left ventricle geometry assessed by left ventricle mass index and relative wall thickness.

CONTACTS AND LOCATIONS:
Overall Officials: Yury A Vasyuk, MD, Principal Investigator — Russian HFS
Locations (1):
- City Hospital №5, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No